CLINICAL TRIAL: NCT01436123
Title: Plasmonic Photothermal and Stem Cell Therapy of Atherosclerosis With The Use of Gold Nanoparticles With Iron Oxide-Silica Shells Versus Stenting
Brief Title: Plasmonic Photothermal and Stem Cell Therapy of Atherosclerosis Versus Stenting
Acronym: NANOM PCI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated under the political pressure of the Federal Security Service of the Russian Federation (FSB) and the Russian Society of Cardiology
Sponsor: Ural State Medical University (Other)
Collaborators: Ural Institute of Cardiology (Other); De Haar Research Foundation (Other); Ural Federal University (Other)
Responsible Party: Principal Investigator, Alexander Kharlamov, Research manager, Ural State Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NANOM PCI
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Plasmonic Photothermal Therapy; Nanoparticles; Stem cells; Atherosclerosis; Bioengineering; Biodegradable stenting; Repair disease
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis | interventions — Stents; Bioengineering

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stenting + Micro-infusion (Experimental): Step 1 - implantation of everolimus-eluting stent with imaging by MSCT, IVUS and OCT; Step 2 - injection of stem cells containing gold nanoparticles with silica-iron oxide shells.
  Interventions: Other: Stenting and micro-infusion of NP
- Stenting (Active Comparator): Put in everolimus-eluting stent
  Interventions: Device: Implantation of everolimus-eluting stent

INTERVENTIONS:
Other: Stenting and micro-infusion of NP — Step 1 - IVUS, OCT-guided put in everolimus-eluting (drug-eluting-DES) stent + intravascular ultrasound (IVUS) mapping + harvesting stem cells with mesenchymal phenotype; Step 2 - culturing of stem cells in medium by gold nanoparticles with silica-iron oxide shells; Step 3 - micro-infusion of stem cells bearing NP into the lesion; Step 4 - detonation of nanoshells after migration of stem cells with NPs inside (until 7-10 days after transplantation). We expect 'melting' and 'burning' effects of PPTT, beneficial effects of bioactive products of stem cells lysis + benefits from further migration of stem cells from patch into the plaque
  Other Names: Plasmonic Photothermal Therapy (PPTT); Stem cell therapy; Bioengineering; Stenting; Xience V stent
  Arms: Stenting + Micro-infusion
Device: Implantation of everolimus-eluting stent — Put stent in ischemia-related coronary artery by indications for PCI
  Other Names: Stenting; Xience V stent
  Arms: Stenting

SUMMARY:
Intensive therapy with rosuvastatin 40 mg and ApoA-I Milano reduces the total atheroma volume (TAV) up to 6.38 or 14.1 mm3 respectively. Our previous bench studies PLASMONICS and NANOM First-in-Man trial documented TAV reduction up to unprecedented 79.4 and 60.3 mm3 respectively with high level of safety and feasibility.

The completed randomized two arm (1:1) study (NANOM-PCI) with parallel assignment (n=62) assessed (NCT01436123) the safety and feasibility of the delivery technique for nanoparticles (NP) using micro-injection catheter (with intravascular intramural injection of allogeneous stem cells carrying NP after MSCT-, IVUS- and OCT-guided mapping of the vessel), and plasmonic photothermal therapy of atherosclerosis combined with stenting (Nano group, n=32) versus stenting with Xience V cage (Stenting group, n=30). The primary outcome was TAV at 12 months.

The mean reduction of TAV at 12 months in Nano group was -84.1 mm3 (95% CI: SD 28.3; min -52.4 mm3, max -99.1 mm3; p<0.05) versus +12.4 mm3 in case of stenting (p<0.05 between groups). 42/62 patients (68%) in Nano group passed the Glagov threshold of a 40% plaque burden with mean plaque burden (PB) 36.2% (95% CI: SD 9.3%, min 30.9%, max 44.5%). The increase of the minimal lumen diameter was 61.2 and 63.3% at 12 month follow up in groups respectively. The serial assessment of VH-IVUS showed a significant decrease at 12 months in the dense calcium area, fibrous and fibro-fatty tissue with fulminant necrosis due to thermolysis in Nano-group, whereas an increase of fibrous and fibro-fatty components in stenting arm. We have documented 2 vs 3 cases of the definite thrombosis and 3 vs 5 cases of target lesion revascularization in groups respectively. The analysis of the event-free survival of the ongoing clinical follow-up shows the significantly lower risk of cardiovascular death in Nano group if compare with conventional stenting (93.4% vs 86.7%; p<0.05).

Plasmonic resonance-mediated therapy using noble-metal NP associated with significant regression of coronary atherosclerosis. Tested delivery approach has acceptable safety and efficacy for atheroregression below a 40% PB.

The investigators hypothesize that multistep approach with the use of stent in acute care unit, and then subsequent transcatheter micro-injection with nanoparticles can resolve atherosclerosis, stop and regress atherogenesis, remodulate or even rejuvenate arteries. Stem cells in patch can be good carriers for nanoparticles as well as high-effective metabolic vectors (paracrine-like regulation of alive cells and via bioactive products of cell lysis after detonation of nanoparticles) for the treatment of plaque on site. Gold nanoparticles with silica-iron oxide shells promise high-energy plasmonic photothermic burning or melting effect under the near-infrared laser irradiation onto the lesion. Thus the investigators expect complex two-side effect on the plaque with protected lumen and adventitia.

Novel discoveries in atherogenesis, and development of nanobiotechnologies with potentials for the management of atherosclerosis leads us to the quest of new approaches. The investigators still cannot really effectively treat atherosclerosis.

The investigators management is more symptomatic, and lipid-pool or inflammation-oriented! The investigators cannot manage non-organic part (mineral deposits, calcified necrotic core, partially collagen and fibrotic tissue) and total plaque volume Surgery and invasive procedures is just focused on blood flow restoration (just manipulate the form of plaque) + concerns of clinical and technical restrictions (incl. alien body - stent) + risk of restenosis or subacute 'fatal' in-stent atherothrombosis + graft survival/ occlusion + surgery-related complications High rate of short- and long-term complications and readmissions. Regression of atherosclerosis in fact is still a dream. The investigators offer an alternative to stenting and may be cardiac artery bypass surgery (CABG). Our approach can really allow to rejuvenate arteries, Plasmonic photothermal therapy (PPTT) can burn plaque, but stem cells and bioengineered structures promise restoration of the vessel wall.

Our personal previous data showed that PPTT can 1.6-fold reduce a volume of plaque with most optimal long-term result in subsets with the use of SPCs as a delivery approach. The most optimal delivery systems of NPs into the plaque are the on-artery bioengineered patch and ferro-magnetic approach.

DETAILED DESCRIPTION:
Nanoparticles (NPs) are quite safe for an organism but entire kinetics is mostly unknown. The most dangerous approach with lowest level of efficacy and safety is a delivery of NPs with microbubbles. SP+ and mesenchymal SPCs have the similar efficacy as a local delivery system with a lot of beneficial properties such as anti-inflammative, anti-apoptotic, and multi-metabolic effects leading to the plaque degradation and artery rejuvenation. Thus, nanoburning is very challenging technique to demolish and reverse the plaque especially in combination with stem cell technologies promising functional restoration of the vessel wall and can be an alternative to stenting.

Altering general strategy the investigators generally offer:

1. The investigators don't need a therapy only with harvested stem cells (not so effective, but more provocative); the investigators have to manage host resident stem cells on site [local in-artery infusion] with growth factors, cytokines [or systemic potentiation, but risk of side effects and adverse events is high].
2. Regular intravenous systemic therapy with modified BM (bone marrow), circulating progenitor, and iPS (induced pluripotent) stem cells might be beneficial for prevention of diseases, and rejuvenation of tissues and organs - but the system as whole will be compromised [the investigators can store stem cells of each individual to use for cell therapy or bioengineering].
3. The best way - development of bioengineered constructions through life to transplant a bioartificial organ on request.
4. Multi-step invasive treatment of atherosclerosis - (1) biodegradable stenting in ACU (acute care unit), or preventively, with no restenosis and no acute atherothrombosis risk profile, (2) regular systemic or local stem cell therapy, or with cytokines, (3) on-artery MSCs (mesenchymal stem cells)-related bioengineered patch with silica-gold iron-bearing NPs [SCs (stem cells) as carriers for NPs with transduction in hands of magnetic fields for local elimination of plaque, and subsequent rejuvenation of artery wall.

Our new approach, challenging modern therapy of atherosclerosis include:

1. BIODEGRADABLE STENTS - for 6-24 months period under the soft short-term antithrombotic therapy (resolving concerns with stenosis/ lumen + steered remodeling); no hemorrhages, no alien metal body, no concerns with further CABG, minimal inflammation
2. INTRAVENOUS NON-SPECIFIC SYSTEMIC STEM CELL THERAPY - before and after stenting - launch repair effects in vessel + beneficial effects for ischemic or injured tissues
3. ON-ARTERY BIOENGINEERED PATCH transplantation with NPs or MICRO-INFUSION of stem cells bearing NP - grown with MSCs and NPs (bovine pericardium scaffold); 3-6 weeks to grow a thin structure (recover cells before or during stenting), multi-effects due to migration of SCs + bioactive products of lysis
4. PLASMONIC PHOTOTHERMAL THERAPY - 'melting' and 'burning' effects - direct degradation + bioactive products of stem cells' lysis + further migration of SCs from patch

Potential expected disadvantages of our approach: Necessity of the special precise delivery technique. Lost function of artery - irreparable pro-fibrotic and pro-inflammative damage - necessity of another clinical approach for restoration of tissue (may be with stem cells). Threat of acute fatal atherothrombosis due to rupture of (vulnerable) plaque - verification of the optimal antithrombotic therapy. Cannot treat non-organic part of plaque - necessity of the special therapy for mineral deposits, calcified necrotic core, fibrotic sites - solution using stem cells. Harm of potent detrimental adverse effects - vapor bubbling (boiling of cytoplasm and ECM with subsequent lysis of cells, and provocation of pro-apoptotic cascades), acoustic and shock waves due to plasma-generated laser-related detonation of nanoshells in tissue - need regenerative therapy (type of SCs, conditions and way of transplantation; Culturing? Sorting?). Erratic (unsteered) heating - surrounding tissue of the site of interest can achieve a temperature until 38-39°. But at the site of burning final temperature can be at about 50-180 C (cauterization/ searing/ melting effect) with consequent pro-fibrotic effect - need regenerative therapy and clarification of energy options.

ELIGIBILITY:
Inclusion Criteria:

* Multivessel coronary artery disease without indications for CABG
* Stable angina with indications for preventive PCI
* NSTEMI (primary PCI and late comers) <=> 12 hr
* STEMI with kept EF>50% (all comers)
* Rescue PCI
* Vessel size between 2.3-4.0 mm
* NYHA II-III functional class of HF
* De novo treatment = no history of PCI or CABG
* Atherosclerosis of proximal left anterior descending artery <50% stenosis
* Treated hypertension
* Signed written informed consent

Exclusion Criteria:

* History of MI
* History of CABG or PCI
* Indications for CABG
* Contraindications for CABG, PCI
* History of unstable angina, coronary artery syndrome
* History of arrhythmias
* History of stroke
* NYHA I, IV functional class of HF
* Diabetes (fasting glucose > 7.0 mM/L)
* Untreated hypertension
* Asthma
* Participation to any drug-investigations during previous 60 days
* Pregnancy
* Intolerance to any limus drugs, aspirin, clopidogrel, aspirin, metals and polymers of stent and nanoparticles
* Need for chronic treatment with anti-vitamin K drugs
* Impossibility of clinical follow-up

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-12; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Total atheroma volume | at month 12
  Total plaque volume measured by intravascular ultrasound (IVUS), cubic mm.

SECONDARY OUTCOMES:
Composite end-point of any MACE (major acute cardiovascular events), all-cause death, any revascularization | at month 12
  Composite end-point of all-cause death, all MACE - major cardiovascular events, any revascularization
Composition of plaque | at month 12
  Analysis of IVUS(intravascular ultrasound)-related composition of plaque (calcified deposits, necrotic calcified core), fibro-lipid core and etc.
Major and minor bleeding | at month 12
  Clinical examination of major and minor bleeding under the antithrombotic therapy
Restenosis rate | at month 12
  Restenosis rate verified clinically + IVUS
Stent thrombosis rate | at month 12
  Stent thrombosis rate verified clinically, angiography, IVUS
Coronary flow-mediated vasodilatation | at month 12
  Ultrasound-related examination of coronary flow-mediated vasodilatation
Coronary intima-media thickness | at month 12
  Ultrasound-IVUS-related examination of coronary intima-media thickness
Minimum diameter stenosis | at month 12
  IVUS-related assessment of minimum diameter stenosis
Minimum lumen diameter | at month 12
  IVUS-related assessment of minimum lumen diameter

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kharlamov, M.D., Ph.D., Principal Investigator — Ural Institute of Cardiology; Jan Gabinsky, M.D., Ph.D., Study Chair — Ural Institute of Cardiology; Olga Kovtun, M.D., Ph.D., Study Director — Ural State Medical University
Locations (3):
- De Haar Research Foundation, Rotterdam, South Holland, Netherlands
- Russia (2):
  - Ural Center of Modern Nanotechnologies, Institute of Natural Sciences, Ural Federal University, Yekaterinburg, Sverdlovsk Oblast
  - Ural Institute of Cardiology, Yekaterinburg, Sverdlovsk Oblast

REFERENCES:
- [Background] Kharlamov AN. Plasmonic photothermal therapy for atheroregression below Glagov threshold. Future Cardiol. 2013 May;9(3):405-25. doi: 10.2217/fca.13.16. PMID 23668744
- See also: Ural Institute of Cardiology — http://www.cardio-burg.ru
- See also: Nanocenter of the Ural Federal University — http://nanocenter.urfu.ru